CLINICAL TRIAL: NCT04204798
Title: Impact of Low-dose Dexmedetomidine on Outcomes of Elderly Admitted to ICU After Noncardiac Surgery: a Randomized Controlled Trial
Brief Title: Dexmedetomidine and Outcomes of Elderly Admitted to ICU After Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University Third Hospital (Other); Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019-226
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Elderly; Surgery; Intensive Care Unit; Dexmedetomidine; Overall Survival
Keywords: Elderly; Surgery; Intensive Care Unit; Dexmedetomidine; Overall survival
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): Dexmedetomidine is infused from 4 pm to 8 am during ICU stay for no more than 3 days.
  Interventions: Drug: Dexmedetomidine
- Placebo group (Placebo Comparator): Normal saline is infused for the same duration as in the dexmedetomidine group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — 1. Dexmedetomidine is infused from 4 pm to 8 am during ICU stay for no more than 3 days.
  2. For non-intubated patients, the infusion rate is adjusted to reach a Richmond Agitation-Sedation Scale (RASS) of -1, or a maximal rate of 0.2 microgram/kg/h, or the occurrence of any adverse events.
  3. For intubated patients, the infusion rate is adjusted to reach a RASS of -1, or a maximal rate of 0.7 microgram/kg/h, or the occurrence of any adverse events.
  Arms: Dexmedetomidine group
Drug: Placebo — 1. Normal saline is infused in the same rate for the same duration as in the dexmedetomidine group.
  2. Propofol sedation is administered when considered necessary.
  Other Names: Normal saline
  Arms: Placebo group

SUMMARY:
Sleep disorder and delirium are common problems in intensive care unit (ICU) patients, and may lead to poor prognosis. The investigators' previous study showed that nighttime infusion of low-dose dexmedetomidine improved the sleep quality and decreased the incidence of delirium in ICU patients after surgery. Long-term follow-up of these patients showed that low-dose dexmedetomidine also improved 2-year survival and the quality of life in 3-year survivors. The purpose of this study is to investigate the effect of low-dose dexmedetomidine on the long-term outcome of elderly patients admitted to the ICU after noncardiac surgery.

DETAILED DESCRIPTION:
Dexmedetomidine is a highly selective α2-adrenoceptor agonist with sedative, analgesic and anti-anxiety properties. Unlike other sedative agents, dexmedetomidine exerts its sedative effects through an endogenous sleep-promoting pathway, producing a state like non-rapid eye movement sleep. For mechanically ventilated patients, sedative-dose dexmedetomidine infusion at night maintains circadian rhythm, increases sleep efficiency, and improves sleep architecture. When used for sedation in mechanical ventilated patients, it reduces the incidence of delirium.

Dexmedetomidine may improve patient outcomes by improving sleep quality. A previous randomized trial found that, for elderly patients who were admitted to ICU after noncardiac surgery, nighttime infusion of low-dose dexmedetomidine significantly improves the sleep quality and decreases the incidence of postoperative delirium. A long-term follow-up of these patients showed that low-dose dexmedetomidine infusion significantly increased survival up to 2 years, and improved cognitive function and quality of life in 3-year survivors.

In the study mentioned above, dexmedetomidine was only infused during the night after surgery with a fixed dose. The investigators hypothesize that, for elderly admitted to ICU after surgery, nighttime infusion of individualized low-dose dexmedetomidine may improve long-term outcomes. This randomized controlled trial is designed to investigate the effect of low-dose dexmedetomidine on 1-year survival and the quality of life of 1-year survivors in elderly patients admitted to the ICU after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years old;
* Admitted to intensive care unit (ICU) after noncardiac surgery;
* Expected to stay in ICU until the next morning. For those with endotracheal intubation, the expected duration of mechanical ventilation is <24 hours;
* Provide written informed consents.

Exclusion Criteria:

* Preoperative history of schizophrenia, epilepsy, Parkinsonism, or myasthenia gravis;
* Inability to communicate in the preoperative period (coma, profound dementia, or language barrier);
* Preoperative history of sleep apnea (previous diagnosis; or STOP-Bang score ≥3 with serum bicarbonate ≥ 28 mmol/L);
* Known sick sinus syndrome, severe sinus bradycardia (<50 beats per min [bpm]), or second degree or higher atrioventricular block without pacemaker;
* Hypotension (systolic blood pressure [SBP] <90 mmHg, mean arterial pressure [MAP] <70 mmHg, or a decrease of SBP >30% of baseline) or in a state of shock (vasopressors are required to maintain MAP ≥65 mmHg and serum lactate >2 mmol/L);
* Severe hepatic dysfunction (Child-Pugh class C), renal failure (requirement of renal replacement therapy), or expected survival <24 hours;
* Traumatic brain injury or neurosurgery;
* Presence of delirium before surgery (assessed with Confusion Assessment Method [CAM]/CAM-ICU);
* Undergoing treatment of dexmedetomidine or clonidine;
* Other conditions that are considered unsuitable for study participation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1410 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2026-06-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival after surgery | Up to 4 years after surgery
  Overall survival after surgery

SECONDARY OUTCOMES:
The incidence of organ injury within 5 days after surgery | Up to 5 days after surgery
  Organ injury include delirium (assessed with Confusion Assessment Method/CAM for the Intensive Care Unit), acute kidney injury (assessed with KIDGO criteria), and myocardial injury (assessed with cardiac troponin I).
Length of stay in the intensive care unit (ICU) stay after surgery | Up to 30 days after surgery
  Length of ICU stay after surgery
Length of stay in hospital after surgery | Up to 30 days after surgery
  Length of stay in hospital after surgery
Incidence of postoperative complications within 30 days after surgery | Up to 30 days after surgery
  Postoperative complications are defined as newly occured medical events that are harmful to patients' recovery and required interventional therapy.
Rate of all-cause 30-day mortality after surgery | Up to 30 days after surgery
  All-cause 30-day mortality after surgery
Sleep quality at 30 days after surgery | At 30 days after surgery
  The sleep quality is assessed with the Pittsburgh Sleep Quality Index Questionnaire (PSQI, score ranges from 0 to 21, with higher score indicating poorer sleep quality).
Recurrence-free survival after surgery | Up to 4 year after surgery
  Recurrence-free survival after surgery
Event-free survival after surgery | Up to 4 year after surgery
  Event-free survival after surgery
Cancer-specific survival after surgery | Up to 4 year after surgery
  Cancer-specific survival after surgery
Quality of life in 1-year survivors after surgery | At the end the 1st year after surgery
  The quality of life is assessed with the World Health Organization Quality of Life Questionaire abbreviated version (WHOQOL-BREF, a 24-item questionnaire that provides assessments of the quality of life in physical, psychological, and social relationship, and environmental domains. For each domain, the score ranges from 0 to 100, with higher score indicating better function).

OTHER OUTCOMES:
Pain severity within 5 days after surgery: Numeric Rating Scale | Up to 5 days after surgery.
  Pain severity is assessed with the Numeric Rating Scale (an 11-point scale where 0=no pain and 10=the worst pain.
Subjective sleep quality within 5 days after surgery: Numeric Rating Scale | Assessed in the morning on the 1st, 2nd, 3rd, 4th, and 5th day after surgery
  Subjective sleep quality the Numeric Rating Scale (an 11-point scale where 0=the best sleep and 10=the worst sleep.
Overall survival after surgery in cancer patients | Up to 4 year after surgery
  Overall survival after surgery in cancer patients
Recurrence-free survival after surgery in cancer patients | Up to 4 year after surgery
  Recurrence-free survival after surgery in cancer patients
Event-free survival after surgery in cancer patients | Up to 4 year after surgery
  Event-free survival after surgery in cancer patients
Cancer-specific survival after surgery in cancer patients | Up to 4 year after surgery
  Cancer-specific survival after surgery in cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Novaes MA, Knobel E, Bork AM, Pavao OF, Nogueira-Martins LA, Ferraz MB. Stressors in ICU: perception of the patient, relatives and health care team. Intensive Care Med. 1999 Dec;25(12):1421-6. doi: 10.1007/s001340051091. PMID 10660851
- [Background] Rotondi AJ, Chelluri L, Sirio C, Mendelsohn A, Schulz R, Belle S, Im K, Donahoe M, Pinsky MR. Patients' recollections of stressful experiences while receiving prolonged mechanical ventilation in an intensive care unit. Crit Care Med. 2002 Apr;30(4):746-52. doi: 10.1097/00003246-200204000-00004. PMID 11940739
- [Background] Simini B. Patients' perceptions of intensive care. Lancet. 1999 Aug 14;354(9178):571-2. doi: 10.1016/S0140-6736(99)02728-2. PMID 10470711
- [Background] Drouot X, Roche-Campo F, Thille AW, Cabello B, Galia F, Margarit L, d'Ortho MP, Brochard L. A new classification for sleep analysis in critically ill patients. Sleep Med. 2012 Jan;13(1):7-14. doi: 10.1016/j.sleep.2011.07.012. Epub 2011 Dec 6. PMID 22153778
- [Background] Gabor JY, Cooper AB, Hanly PJ. Sleep disruption in the intensive care unit. Curr Opin Crit Care. 2001 Feb;7(1):21-7. doi: 10.1097/00075198-200102000-00004. PMID 11373507
- [Background] Freedman NS, Gazendam J, Levan L, Pack AI, Schwab RJ. Abnormal sleep/wake cycles and the effect of environmental noise on sleep disruption in the intensive care unit. Am J Respir Crit Care Med. 2001 Feb;163(2):451-7. doi: 10.1164/ajrccm.163.2.9912128. PMID 11179121
- [Background] Elliott R, McKinley S, Cistulli P, Fien M. Characterisation of sleep in intensive care using 24-hour polysomnography: an observational study. Crit Care. 2013 Mar 18;17(2):R46. doi: 10.1186/cc12565. PMID 23506782
- [Background] Aurell J, Elmqvist D. Sleep in the surgical intensive care unit: continuous polygraphic recording of sleep in nine patients receiving postoperative care. Br Med J (Clin Res Ed). 1985 Apr 6;290(6474):1029-32. doi: 10.1136/bmj.290.6474.1029. PMID 3921096
- [Background] Gabor JY, Cooper AB, Crombach SA, Lee B, Kadikar N, Bettger HE, Hanly PJ. Contribution of the intensive care unit environment to sleep disruption in mechanically ventilated patients and healthy subjects. Am J Respir Crit Care Med. 2003 Mar 1;167(5):708-15. doi: 10.1164/rccm.2201090. PMID 12598213
- [Background] Esquinas AM, Papadakos PJ, Schwartz AR. Sleep patterns during long-term mechanical ventilation in tracheostomized patients in the ICU: do they matter? Crit Care Med. 2014 Jan;42(1):e82-3. doi: 10.1097/CCM.0b013e3182a84ccd. No abstract available. PMID 24346550
- [Background] Day A, Haj-Bakri S, Lubchansky S, Mehta S. Sleep, anxiety and fatigue in family members of patients admitted to the intensive care unit: a questionnaire study. Crit Care. 2013 May 24;17(3):R91. doi: 10.1186/cc12736. PMID 23705988
- [Background] Hu RF, Jiang XY, Zeng YM, Chen XY, Zhang YH. Effects of earplugs and eye masks on nocturnal sleep, melatonin and cortisol in a simulated intensive care unit environment. Crit Care. 2010;14(2):R66. doi: 10.1186/cc8965. Epub 2010 Apr 18. PMID 20398302
- [Background] Kondili E, Alexopoulou C, Xirouchaki N, Georgopoulos D. Effects of propofol on sleep quality in mechanically ventilated critically ill patients: a physiological study. Intensive Care Med. 2012 Oct;38(10):1640-6. doi: 10.1007/s00134-012-2623-z. Epub 2012 Jul 3. PMID 22752356
- [Background] Hardin KA, Seyal M, Stewart T, Bonekat HW. Sleep in critically ill chemically paralyzed patients requiring mechanical ventilation. Chest. 2006 Jun;129(6):1468-77. doi: 10.1378/chest.129.6.1468. PMID 16778263
- [Background] Roberts B, Rickard CM, Rajbhandari D, Turner G, Clarke J, Hill D, Tauschke C, Chaboyer W, Parsons R. Multicentre study of delirium in ICU patients using a simple screening tool. Aust Crit Care. 2005 Feb;18(1):6, 8-9, 11-4 passim. doi: 10.1016/s1036-7314(05)80019-0. PMID 18038529
- [Background] Balas MC, Happ MB, Yang W, Chelluri L, Richmond T. Outcomes Associated With Delirium in Older Patients in Surgical ICUs. Chest. 2009 Jan;135(1):18-25. doi: 10.1378/chest.08-1456. Epub 2008 Nov 18. PMID 19017895
- [Background] Ansaloni L, Catena F, Chattat R, Fortuna D, Franceschi C, Mascitti P, Melotti RM. Risk factors and incidence of postoperative delirium in elderly patients after elective and emergency surgery. Br J Surg. 2010 Feb;97(2):273-80. doi: 10.1002/bjs.6843. PMID 20069607
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Franco K, Litaker D, Locala J, Bronson D. The cost of delirium in the surgical patient. Psychosomatics. 2001 Jan-Feb;42(1):68-73. doi: 10.1176/appi.psy.42.1.68. PMID 11161124
- [Background] Milbrandt EB, Deppen S, Harrison PL, Shintani AK, Speroff T, Stiles RA, Truman B, Bernard GR, Dittus RS, Ely EW. Costs associated with delirium in mechanically ventilated patients. Crit Care Med. 2004 Apr;32(4):955-62. doi: 10.1097/01.ccm.0000119429.16055.92. PMID 15071384
- [Background] Pisani MA, Kong SY, Kasl SV, Murphy TE, Araujo KL, Van Ness PH. Days of delirium are associated with 1-year mortality in an older intensive care unit population. Am J Respir Crit Care Med. 2009 Dec 1;180(11):1092-7. doi: 10.1164/rccm.200904-0537OC. Epub 2009 Sep 10. PMID 19745202
- [Background] Bickel H, Gradinger R, Kochs E, Forstl H. High risk of cognitive and functional decline after postoperative delirium. A three-year prospective study. Dement Geriatr Cogn Disord. 2008;26(1):26-31. doi: 10.1159/000140804. Epub 2008 Jun 24. PMID 18577850
- [Background] Van Rompaey B, Schuurmans MJ, Shortridge-Baggett LM, Truijen S, Elseviers M, Bossaert L. Long term outcome after delirium in the intensive care unit. J Clin Nurs. 2009 Dec;18(23):3349-57. doi: 10.1111/j.1365-2702.2009.02933.x. Epub 2009 Sep 4. PMID 19735334
- [Background] Salas RE, Gamaldo CE. Adverse effects of sleep deprivation in the ICU. Crit Care Clin. 2008 Jul;24(3):461-76, v-vi. doi: 10.1016/j.ccc.2008.02.006. PMID 18538195
- [Background] Kamdar BB, Needham DM, Collop NA. Sleep deprivation in critical illness: its role in physical and psychological recovery. J Intensive Care Med. 2012 Mar-Apr;27(2):97-111. doi: 10.1177/0885066610394322. Epub 2011 Jan 10. PMID 21220271
- [Background] Patel J, Baldwin J, Bunting P, Laha S. The effect of a multicomponent multidisciplinary bundle of interventions on sleep and delirium in medical and surgical intensive care patients. Anaesthesia. 2014 Jun;69(6):540-9. doi: 10.1111/anae.12638. PMID 24813132
- [Background] Hu RF, Jiang XY, Chen J, Zeng Z, Chen XY, Li Y, Huining X, Evans DJ. Non-pharmacological interventions for sleep promotion in the intensive care unit. Cochrane Database Syst Rev. 2015 Oct 6;2015(10):CD008808. doi: 10.1002/14651858.CD008808.pub2. PMID 26439374
- [Background] Chen CJ, Hsu LN, McHugh G, Campbell M, Tzeng YL. Predictors of sleep quality and successful weaning from mechanical ventilation among patients in respiratory care centers. J Nurs Res. 2015 Mar;23(1):65-74. doi: 10.1097/jnr.0000000000000066. PMID 25668737
- [Background] Knill RL, Moote CA, Skinner MI, Rose EA. Anesthesia with abdominal surgery leads to intense REM sleep during the first postoperative week. Anesthesiology. 1990 Jul;73(1):52-61. doi: 10.1097/00000542-199007000-00009. PMID 2360740
- [Background] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Background] Cooper AB, Thornley KS, Young GB, Slutsky AS, Stewart TE, Hanly PJ. Sleep in critically ill patients requiring mechanical ventilation. Chest. 2000 Mar;117(3):809-18. doi: 10.1378/chest.117.3.809. PMID 10713011
- [Background] Rosenberg-Adamsen S, Skarbye M, Wildschiodtz G, Kehlet H, Rosenberg J. Sleep after laparoscopic cholecystectomy. Br J Anaesth. 1996 Nov;77(5):572-5. doi: 10.1093/bja/77.5.572. PMID 8957969
- [Background] Pisani MA, Friese RS, Gehlbach BK, Schwab RJ, Weinhouse GL, Jones SF. Sleep in the intensive care unit. Am J Respir Crit Care Med. 2015 Apr 1;191(7):731-8. doi: 10.1164/rccm.201411-2099CI. PMID 25594808
- [Background] Kanji S, Mera A, Hutton B, Burry L, Rosenberg E, MacDonald E, Luks V. Pharmacological interventions to improve sleep in hospitalised adults: a systematic review. BMJ Open. 2016 Jul 29;6(7):e012108. doi: 10.1136/bmjopen-2016-012108. PMID 27473952
- [Background] Krenk L, Jennum P, Kehlet H. Postoperative sleep disturbances after zolpidem treatment in fast-track hip and knee replacement. J Clin Sleep Med. 2014 Mar 15;10(3):321-6. doi: 10.5664/jcsm.3540. PMID 24634631
- [Background] Kishi T, Matsunaga S, Iwata N. Suvorexant for Primary Insomnia: A Systematic Review and Meta-Analysis of Randomized Placebo-Controlled Trials. PLoS One. 2015 Aug 28;10(8):e0136910. doi: 10.1371/journal.pone.0136910. eCollection 2015. PMID 26317363
- [Background] Mo Y, Scheer CE, Abdallah GT. Emerging Role of Melatonin and Melatonin Receptor Agonists in Sleep and Delirium in Intensive Care Unit Patients. J Intensive Care Med. 2016 Aug;31(7):451-5. doi: 10.1177/0885066615592348. Epub 2015 Jun 19. PMID 26092575
- [Background] Akeju O, Hobbs LE, Gao L, Burns SM, Pavone KJ, Plummer GS, Walsh EC, Houle TT, Kim SE, Bianchi MT, Ellenbogen JM, Brown EN. Dexmedetomidine promotes biomimetic non-rapid eye movement stage 3 sleep in humans: A pilot study. Clin Neurophysiol. 2018 Jan;129(1):69-78. doi: 10.1016/j.clinph.2017.10.005. Epub 2017 Oct 20. PMID 29154132
- [Background] Alexopoulou C, Kondili E, Diamantaki E, Psarologakis C, Kokkini S, Bolaki M, Georgopoulos D. Effects of dexmedetomidine on sleep quality in critically ill patients: a pilot study. Anesthesiology. 2014 Oct;121(4):801-7. doi: 10.1097/ALN.0000000000000361. PMID 24988068
- [Background] Nelson LE, Lu J, Guo T, Saper CB, Franks NP, Maze M. The alpha2-adrenoceptor agonist dexmedetomidine converges on an endogenous sleep-promoting pathway to exert its sedative effects. Anesthesiology. 2003 Feb;98(2):428-36. doi: 10.1097/00000542-200302000-00024. PMID 12552203
- [Background] Goettel N, Bharadwaj S, Venkatraghavan L, Mehta J, Bernstein M, Manninen PH. Dexmedetomidine vs propofol-remifentanil conscious sedation for awake craniotomy: a prospective randomized controlled trial. Br J Anaesth. 2016 Jun;116(6):811-21. doi: 10.1093/bja/aew024. Epub 2016 Apr 20. PMID 27099154
- [Background] Lu Z, Li W, Chen H, Qian Y. Efficacy of a Dexmedetomidine-Remifentanil Combination Compared with a Midazolam-Remifentanil Combination for Conscious Sedation During Therapeutic Endoscopic Retrograde Cholangio-Pancreatography: A Prospective, Randomized, Single-Blinded Preliminary Trial. Dig Dis Sci. 2018 Jun;63(6):1633-1640. doi: 10.1007/s10620-018-5034-3. Epub 2018 Mar 29. PMID 29594976
- [Background] Silva-Jr JM, Katayama HT, Nogueira FAM, Moura TB, Alves TL, de Oliveira BW. Comparison of dexmedetomidine and benzodiazepine for intraoperative sedation in elderly patients: a randomized clinical trial. Reg Anesth Pain Med. 2019 Mar;44(3):319-324. doi: 10.1136/rapm-2018-100120. Epub 2019 Feb 3. PMID 30777901
- [Background] Wu XH, Cui F, Zhang C, Meng ZT, Wang DX, Ma J, Wang GF, Zhu SN, Ma D. Low-dose Dexmedetomidine Improves Sleep Quality Pattern in Elderly Patients after Noncardiac Surgery in the Intensive Care Unit: A Pilot Randomized Controlled Trial. Anesthesiology. 2016 Nov;125(5):979-991. doi: 10.1097/ALN.0000000000001325. PMID 27571256
- [Background] Riker RR, Shehabi Y, Bokesch PM, Ceraso D, Wisemandle W, Koura F, Whitten P, Margolis BD, Byrne DW, Ely EW, Rocha MG; SEDCOM (Safety and Efficacy of Dexmedetomidine Compared With Midazolam) Study Group. Dexmedetomidine vs midazolam for sedation of critically ill patients: a randomized trial. JAMA. 2009 Feb 4;301(5):489-99. doi: 10.1001/jama.2009.56. Epub 2009 Feb 2. PMID 19188334
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303